CLINICAL TRIAL: NCT00563303
Title: Interest of Treatment of Polytraumatisms With Corticoids (Hydrocortisone) for Patient With Relative Adrenocortical Insufficiency
Brief Title: Treatment of Polytraumatisms With Corticoids
Acronym: Hypolyte
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Serb (Unknown)
Responsible Party: Pierre-joachim Mahé, investigator coordinator, CHu de Nantes
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BRD 06/6-L; Afssaps: 060785; CPP: 2006/25
Record Dates: First submitted 2006-09-26; First posted 2007-11-26 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Polytraumatism
MeSH Terms: conditions — Multiple Trauma | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- H (Experimental): Hydrocortisone
  Interventions: Drug: hydrocortisone
- P (Placebo Comparator): Treatment by NaCl (placebo)
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: hydrocortisone — 200mg/jour (solution of 48mL), Day 1 to Day 4 100mg/jour (solution of 48mL), Day 5 50mg/jour (solution of 48mL), Day 6
  Arms: H
Drug: NaCl — 48mL from Day 1 to Day 6
  Arms: P

SUMMARY:
Interest of treatment of polytraumatisms with corticoids (hydrocortisone) for patient with relative adrenocortical insufficiency on frequency of nosocomial infection, and hemodynamic complications and organs injuries.

ELIGIBILITY:
Inclusion Criteria:

* Age superior of 15 years
* Hospitalization in reanimation for polytraumatism (lesion of two organs with a vital risk)
* SISS score more than 15
* Intubation for more than 48 hours.
* Agreement of a family member
* Patient with insurance

Exclusion Criteria:

* History of corticothérapies within 6 months
* History of adrenocortical insufficiency.
* Treatment by immunosuppressor
* Immunodeficiency.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-11; Primary Completion 2006-11 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Incidence of nosocomial pneumopathy: radiological, clinical and bacteriological criteria | 28 days

SECONDARY OUTCOMES:
Incidence of bacteremia, urinary infections, infections of the operatory sites, incidence of SDRA, organ dysfunction,mortality, etc. | 28 days
Incidence of nosocomial pneumopathy | Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Mahe Joachim, MD, Principal Investigator — Nantes University Hospital
Locations (7):
- France (7):
  - CHU Bordeaux, Bordeaux
  - CHU Morvan de Brest, Brest
  - CHU Caen, Caen
  - CH La Roche Sur Yon, La Roche-sur-Yon
  - Hôtel Dieu, Nantes
  - CHU Pontchaillou, Rennes
  - CHU Trousseau, Tours

REFERENCES:
- [Derived] Le Bras M, Roquilly A, Deckert V, Langhi C, Feuillet F, Sebille V, Mahe PJ, Bach K, Masson D, Lagrost L, Costet P, Asehnoune K, Cariou B. Plasma PCSK9 is a late biomarker of severity in patients with severe trauma injury. J Clin Endocrinol Metab. 2013 Apr;98(4):E732-6. doi: 10.1210/jc.2012-4236. Epub 2013 Feb 28. PMID 23450051
- [Derived] Asehnoune K, Mahe PJ, Seguin P, Jaber S, Jung B, Guitton C, Chatel-Josse N, Subileau A, Tellier AC, Masson F, Renard B, Malledant Y, Lejus C, Volteau C, Sebille V, Roquilly A. Etomidate increases susceptibility to pneumonia in trauma patients. Intensive Care Med. 2012 Oct;38(10):1673-82. doi: 10.1007/s00134-012-2619-8. Epub 2012 Jul 10. PMID 22777514
- [Derived] Roquilly A, Mahe PJ, Seguin P, Guitton C, Floch H, Tellier AC, Merson L, Renard B, Malledant Y, Flet L, Sebille V, Volteau C, Masson D, Nguyen JM, Lejus C, Asehnoune K. Hydrocortisone therapy for patients with multiple trauma: the randomized controlled HYPOLYTE study. JAMA. 2011 Mar 23;305(12):1201-9. doi: 10.1001/jama.2011.360. PMID 21427372